CLINICAL TRIAL: NCT04481451
Title: Quadratus Lumborum vs Erector Spinae Supplementary Blocks With Lumbar Plexus Blocks for Hip PAO
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of interest.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Roland Brusseau, Director, Pediatric Regional Anesthesia Services, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-P00034474
Record Dates: First submitted 2020-07-15; First posted 2020-07-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative; Regional Anesthesia; Hip Dysplasia
Keywords: pain; regional anesthesia; regional block; lumbar plexus block; erector spinae block; paravertebral block; continuous nerve block; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Hip Dislocation; Pain | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: 2 arm randomized controlled non-inferiority trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The identity of the study block type will be hidden from caregivers unless clinically mandated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Erector spinae supplemental block (Experimental): Single-shot T9/T10 operative side erector spinae block using ropivacaine 0.2%, 0.5ml/kg.
  Interventions: Procedure: Erector spinae block with ropivacaine 0.2%; Drug: Ropivacaine
- Quadratus lumborum supplemental block (Active Comparator): Single-shot T9/T10 operative side quadratus lumborum (type 1) block using ropivacaine 0.2%, 0.5ml/kg.
  Interventions: Procedure: Quadratus lumborum block with ropivacaine 0.2%; Drug: Ropivacaine

INTERVENTIONS:
Procedure: Erector spinae block with ropivacaine 0.2% — Single-shot ultrasound-guided nerve block performed ipsilateral to surgical site.
  Other Names: regional nerve block; ropivacaine
  Arms: Erector spinae supplemental block
Procedure: Quadratus lumborum block with ropivacaine 0.2% — Single-shot ultrasound-guided nerve block performed ipsilateral to surgical site.
  Other Names: regional nerve block; ropivacaine
  Arms: Quadratus lumborum supplemental block
Drug: Ropivacaine — ropivacaine 0.2% nerve block injection
  Other Names: Naropin

SUMMARY:
This study proposes to evaluate the efficacy of single shot erector spinae block (ESB) versus single shot quadratus lumborum block (QLB) when used in conjunction with continuous lumbar plexus block (LPB) for postoperative analgesia in children and adolescents undergoing unilateral hip surgical procedures. The aim of this study is to compare the efficacy of the QL vs. ESP blocks as supplements to the lumbar plexus block with respect to pain control outcomes after hip PAO surgery. Both blocks are safe and easy to perform. There is currently no comparative, prospective data concerning the use of these two blocks for hip surgery. The investigational hypothesis is that there will be no clinical difference in the amount of opioid consumed or the overall pain control offered by these two block options.

DETAILED DESCRIPTION:
The Bernese periacetabular osteotomy (PAO) is currently performed at this institution as a non-arthroplasty option to treat developmental hip dysplasia in symptomatic adolescents and young adults. Extensive orthopedic surgical procedures of the hip such as this are associated with severe postoperative pain and benefit from regional anesthesia which provides dense, targeted analgesia to selected dermatomes. These blocks have the potential to decrease opioid exposure intraoperatively and postoperatively, thus avoiding opioid-related side effects such as nausea and vomiting. Other well-known benefits of regional anesthesia in other surgeries include earlier extubation, shorter ICU admissions, shortened post anesthesia care unit (PACU) stays, earlier mobilization, facilitation of physical therapy, improving patient satisfaction, and improved comfort during recovery process. The opioid sparing advantages of regional anesthesia are particularly relevant given the current concerns over the opioid epidemic and data relating opioid administration around surgery recovery and long-term opioid use.

Innervation of the hip is very complex with contributions from various neural structures arising from the lumbar plexus, including branches of the femoral nerve (L2-L4) innervating the anterolateral capsule and obturator nerve (L2-L4) innervating the anteromedial capsule. The posterior and inferior part of the hip joint are innervated by the sacral plexus consisting of the superior gluteal nerve (L4-S1) and branches of the sciatic (L4-S3) including the nerve to rectus femoris (L4-S1).

The skin areas involved in the two most common hip PAO surgery incisions (ilioinguinal incision or the iliofemoral incision) include territories that are innervated by subcostal nerve (T12) and ilioinguinal and iliohypogastric nerves (L1), 4 neural structures not reliably covered with the lumbar plexus block given their origin far more superior from the point of injection which is usually between L2 and L4. For this reason, supplemental blocks such as the ESB and QLB have been employed to improve nerve block coverage and pain control. The lateral femoral cutaneous nerve (L1) which is a sensory branch of the lumbar plexus that supplies skin of the lateral thigh, has a less important role in this context given that the surgical incisions are far more anterior to its territory of innervation.

Surgical osteotomies commonly associated with the Bernese procedure are performed on the anterior portion of the ischium, superior pubic ramus, posterior; partial osteotomies of the ischium below the acetabulum are common as well. Arthrotomy is only performed in selected cases if there is concern for intraarticular pathology, such as a torn labrum, lesions of the femoral neck, or loose bodies. The pelvic bone with its respective osteotome (i.e. bone) innervation includes territories ranging from L2 to S1.7 Some evidence suggest that the iliac crest receives its main sensory innervation from femoral nerve while the gluteal surface of the ilium comes from the sciatic nerve.

Given the many dermatomes and osteotomes that are involved, various regional anesthetic techniques have been described, including LPB, fascia iliaca block, femoral nerve block, obturator nerve block, sacral plexus block, paravertebral blocks, and also interfascial plane blocks like QLB and ESB.

The lumbar plexus block has been shown to provide prolonged analgesia and reduced analgesic requirements in postoperative period for pediatric patients undergoing hip surgery. This block targets mainly femoral, obturator, and lateral femoral cutaneous nerves. At this institution, ultrasound-guided lumbar plexus block using the "shamrock method" has been performed as standard of care for PAO surgery.

Skin incisions include dermatomes T12 to L1 that are not usually covered by the lumbar plexus block. For full coverage, it is necessary to add a supplementary block to cover these dermatomes. The options for this coverage are the QLB, the ESB, or paravertebral block (PVB). Due to the lack of evidence of superiority for any one of these additional blocks over another, the choice of the block is most often made based on the preference of the regional anesthesia team. All three blocks have been reported as effectively covering the cutaneous incision areas. A retrospective preliminary analysis of local data comparing these supplementary blocks suggested a potential difference favoring ESB in terms of opioid consumption when compared to PV or QL.

The QLB blocks the anterior branches of thoracoabdominal nerves and may extend to the upper branches of the lumbar plexus and lateral cutaneous branches of the thoracoabdominal nerves with possible spread to the paravertebral space. There are at least four different variants described in literature based on the site of injection in relation to the quadratus lumborum muscle: type 1 (lateral), type 2 (posterior), type 3 (anterior or transmuscular) and type 4 (intramuscular) - each causing different spread patterns of injectate with affected dermatomes ranging from thoracic T6 to lumbar L2. There is no literature evidence suggesting that one specific QLB approach is superior than the others in terms of clinical outcomes or duration in this setting.

The ESB is a novel block developed in 2016. A rapidly growing body of literature suggests it is efficacious in relieving back, chest wall, abdominal wall and flank pain in both acute and chronic settings. It has been shown to be a viable option for breast, spine, thoracic and abdominal surgical procedures. Recently it has also been reported as an alternative for hip surgery analgesia. Depending on the level of application, this block permits an extensive craniocaudal spread of the local anesthetic along the fascial plane underlying erector spinae muscle allowing multiple dermatomal coverage from a single injection. At lumbar level it can spread from the T12 to S1 vertebrae.

The aim of our study is to compare the efficacy of the QL vs. ESB blocks as supplements to the lumbar plexus block with respect to pain control outcomes after hip PAO surgery. Both blocks are safe and easy to perform. There is currently no comparative, prospective data concerning the use of these two blocks for hip surgery. The investigational hypothesis is that there will be no clinical difference in the amount of opioid consumed or the overall pain control offered by these two block options.

The investigators propose a randomized, controlled, non-inferiority trial to compare the effectiveness of QLBs versus ESBs as supplementary blocks to continuous LPB for patients undergoing primary periacetabular osteotomies. They will compare rescue analgesic requirements, rendered as opiate equivalents, at 24, 48 and 72 hours postoperatively as the primary endpoint. Patients aged 15 years - 30 years of age will be recruited from the home insitution.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I - III status, undergoing unilateral periacetabular osteotomy for treating primary diagnosis of developmental acetabular dysplasia in symptomatic young patients.
2. Ages 15 - 30 years

Exclusion Criteria:

1. Patients undergoing procedures including revision PAO, bilateral PAO, conversion to total hip arthroplasty.
2. Patients whom for any reason did not received a lumbar plexus catheter as part of the baseline regional anesthesia plan
3. Patients with body mass index (BMI) > 35
4. Patients with known coagulopathies.
5. Patients with severe neurodevelopmental delays.
6. Patients with previous chronic pain syndromes.
7. Patients with a history of opioid treatment at any point in the 2 months prior to surgery.
8. Lack of parental consent and/or patient assent.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Rescue analgesic consumption | Day 1
  Opioid use via PCA

SECONDARY OUTCOMES:
Mean pain scores | Every 12 hours
  Numerical rating scale for pain (0-10, with 10 indicating most pain)
PACU Time | PACU stay
  Total time spent in PACU
Adverse events | 2 weeks
  Any unexpected outcome attributable to intervention

CONTACTS AND LOCATIONS:
Overall Officials: ROLAND BRUSSEAU, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children"S Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No